CLINICAL TRIAL: NCT01114256
Title: FNA Tumor Sampling for CD137 Modulation: A Pilot Study
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: VAR0053; SU-04072010-5602 (Other: Stanford University)
Record Dates: First submitted 2010-04-23; First posted 2010-05-03 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Head and Neck Cancer; Breast Cancer; Head and Neck Cancers; Non-Hodgkin Lymphoma; Colorectal Adenocarcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Breast Neoplasms; Lymphoma, Non-Hodgkin | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood, fine needle aspiration biopsy

GROUPS / COHORTS (1):
- Fine needle aspiration (FNA) biopsies: Fine needle aspiration biopsies (FNA) will be performed prior to and 0 to 336 hours after the therapeutic monoclonal antibody infusion.
  Interventions: Procedure: FNA Biopsy

INTERVENTIONS:
Procedure: FNA Biopsy

SUMMARY:
The purpose of this study is to better understand the biology of the body's immune response to monoclonal antibody therapy for cancer. Your health information will be used to identify your tissues. The tissue we obtain may be useful for research or education, resulting in new drugs, therapies or diagnostic procedures.

ELIGIBILITY:
ALL Patients:

1. Patient must have a lymphoma, squamous cell carcinoma of the head and neck, HER2+ breast adenocarcinoma, colorectal adenocarcinoma, or other solid tumor.
2. Patients must not have received any immunosuppressive or anti cancer agent within 2 weeks prior to the first planned FNA biopsy.
3. The patient's therapeutic plan must include a standard therapeutic monoclonal antibody (such as rituximab, cetuximab/panitumumab or trastuzumab) or an investigational monoclonal antibody) to be administered on a schedule such that a FNA biopsy can be done within one week prior, and/or peripheral blood drawn immediately prior to the first dose of the therapeutic mAb and immediately to 24-336 hours post dose. Patients not receiving any other anti- cancer or immunosuppressive (steroids) modality within that time frame are preferred, though use of such agents does not exclude them from the study.
4. Patients not receiving any immunosuppressive or anti-cancer agent within 2 weeks prior to the first planned FNA biopsy are preferred.
5. Informed consent must occur and be documented per institutional rules prior to the first planned FNA biopsy and blood draw.

Patients Providing an FNA in addition to Blood Samples: Criteria applicable to FNA, and not required for patients providing PBMCs without FNA. Patients without tumors amenable to FNA will be candidates for blood sampling only.

If patients do not meet inclusion criteria, then they will be excluded from participating in this study.

1. Patients must have a normal WBC and platelet count, must have no evidence of coagulopathy and must not have received irreversible platelet inhibitors (aspirin) for 2 weeks and reversible platelet inhibitors (other NSAIDS) for one week prior to the initial FNA biopsy.
2. Patients may not be taking therapeutic anticoagulation (target INR of >=2) (warfarin or heparin).
3. Patients must have tumor masses amenable to minimally invasive fine needle aspiration by direct visualization and/ or palpation of the tumor. Generally this will be a biopsy of the primary tumor site or superficial regional lymph nodes.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Stanford Cancer Center with lymphoma, squamous cell carcinoma of the head and neck, HER2+ breast adenocarcinoma, colorectal adenocarcinoma, or other solid tumor.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2010-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
evaluation of change in CD137 positive NK cells in blood & tumors in response to therapeutic moAbs | 12 months

SECONDARY OUTCOMES:
Evaluation of activation status of CD137 positive NK cells | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. A. Dimitrios Colevas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Makkouk A, Sundaram V, Chester C, Chang S, Colevas AD, Sunwoo JB, Maecker H, Desai M, Kohrt HE. Characterizing CD137 upregulation on NK cells in patients receiving monoclonal antibody therapy. Ann Oncol. 2017 Feb 1;28(2):415-420. doi: 10.1093/annonc/mdw570. PMID 27831501